CLINICAL TRIAL: NCT03175523
Title: HOW To Optimally Implant BioResorbable Scaffold - Intravascular Imaging Versus Quantitative Coronary Angiography Guidance
Acronym: HOWTO-BRS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: BioResorbable Scaffold is not available in South Korea
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2017-03
Record Dates: First submitted 2017-05-31; First posted 2017-06-05 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Coronary Stenosis
Keywords: BioResorbable Scaffold; Quantitative Coronary Angiography; Intravascular Imaging
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imaging guided Bioresorbable scaffold (Active Comparator)
  Interventions: Device: imaging guided Bioresorbable scaffold implantation
- QCA-guided Bioresorbable scaffold (Experimental): quantitative coronary angiography guided Bioresorbable scaffold
  Interventions: Device: quantitative coronary angiography guided Bioresorbable scaffold implantation

INTERVENTIONS:
Device: quantitative coronary angiography guided Bioresorbable scaffold implantation — In the QCA-guided group, BRS size and length were chosen by both visual estimation and on-line QCA, and adjunct high-pressure dilation is routinely performed to achieve angiographic residual diameter stenosis less than 30% by QCA and absence of angiographically visible dissections.
  Arms: QCA-guided Bioresorbable scaffold
Device: imaging guided Bioresorbable scaffold implantation — In the imaging-guided group, imaging is used at any step of percutaneous coronary intervention(PCI) before, during, or after PCI. Final image examination after PCI is mandatory.
  Arms: Imaging guided Bioresorbable scaffold

SUMMARY:
The objective of this trial is to compare clinical outcomes between imaging-guided and QCA-guided strategy in patients with native coronary artery disease undergoing BRS implantation.

DETAILED DESCRIPTION:
The investigators hypothesized that intravascular imaging-guided BRS implantation is superior to QCA-guided BRS implantation with respect to target lesion failure in patients with native coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 19 years of age
* Typical chest pain or objective evidence of myocardial ischemia suitable for elective percutaneous coronary intervention
* Native coronary artery lesions with lesion length 50mm and less and reference vessel diameter of 2.5 ~ 3.75mm by quantitative coronary angiography assessment
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

* Angiographic exclusion criteria: any of the followings

  1. Small vessel: mean reference size < 2.5 mm by quantitative coronary angiography
  2. True bifurcation lesion with a large side branch (reference vessel diameter > 2.3mm) requiring a complex two-stent approach
  3. Left main lesions
  4. Ostial lesions within 3mm of the origin: right coronary artery, left anterior descending, or left circumflex artery
  5. Impaired delivery of the Absorb bio- resorbable vascular scaffold is expected:

     * Extreme angulation (≥90°) proximal to or within the target lesion.
     * Excessive tortuosity (≥two 45° angles) proximal to or within the target lesion.
     * Moderate or heavy calcification proximal to or within the target lesion.
  6. In-stent restenotic lesions
* ST-elevation myocardial infarction undergoing primary percutaneous coronary intervention (with 12- 24 hour after symptoms onset)
* Prior percutaneous coronary intervention within the target vessel during the last 12 months.
* Prior percutaneous coronary intervention within the non-target vessel or any peripheral intervention is acceptable if performed anytime >30 days before the index procedure, or between 24 hours and 30 days before the index procedure if successful and uncomplicated.
* Left ventricular ejection fraction (LVEF) < 30%
* Hypersensitivity or contraindication to device material and its degradants (everolimus, poly (L-lactide), poly (DL-lactide), lactide, lactic acid) and cobalt, chromium, nickel, platinum, tungsten, acrylic and fluoro polymers that cannot be adequately pre-medicated.
* Persistent thrombocytopenia (platelet count <100,000/µl)
* Any history of hemorrhagic stroke or intracranial hemorrhage, transient ischemic attack or ischemic stroke within the past 6 months
* A known intolerance to a study drug (aspirin, clopidogrel or ticagrelor)
* Patients requiring long-term oral anticoagulants or cilostazol
* Any surgery requiring general anesthesia or discontinuation of aspirin and/or an Adenosine diphosphate(ADP) antagonist is planned within 12 months after the procedure.
* A diagnosis of cancer (other than superficial squamous or basal cell skin cancer) in the past 3 years or current treatment for the active cancer.
* Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the Investigator, would preclude safe completion of the study.
* Hepatic disease or biliary tract obstruction, or significant hepatic enzyme elevation (alanine transaminase (ALT) or aspartate transaminase (AST) > 3 times upper limit of normal).
* Life expectancy < 5 years for any non-cardiac or cardiac causes
* Unwillingness or inability to comply with the procedures described in this protocol.
* Patient's pregnant or breast-feeding or child-bearing potential.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Target lesion failure | 1 year
  the cumulative incidence of cardiac death, target vessel myocardial infarction or ischemia-driven target lesion revascularization at 12 months after the index procedure.

SECONDARY OUTCOMES:
Device success | 1 hour after an index procedure
  Successful delivery and deployment of the study scaffold at the intended target lesion and successful withdrawal of the delivery system with attainment of final in-scaffold residual stenosis of less than 30% by quantitative coronary angiography (QCA).
Procedural success | 24 hours after an index procedure
  Achievement of final in-scaffold residual stenosis of less than 30% by quantitative coronary angiography with successful delivery and deployment of at least one study scaffold at the intended target lesion and successful withdrawal of the delivery system for all target lesions without the occurrence of cardiac death, target vessel myocardial infarction or repeat target lesion revascularization during the hospital stay.
Death | 1 year, and 5 years
  cardiac, vascular, non-cardiovascular
Myocardial infarction | 1 year, and 5 years
Scaffold thrombosis | 1 year, and 5 years
Stroke | 1 year, and 5 years
Target lesion revascularization | 1 year, and 5 years
Any revascularization | 1 year, and 5 years
Target lesion failure (TLR) | 1 year, and 5 years
  cardiac death, target vessel myocardial infarction or ischemia-driven target lesion revascularization
A composite event | 1 year, and 5 years
  a composite event of cardiac death, target vessel myocardial infarction, stroke, or clinically significant bleeding(clinically significant bleeding by Bleeding Academic Research Consortium (BARC) type 2,3,4,5)
In-scaffold restenosis on coronary CT angiography | 1 year, and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yang-soo Jang, MD, Principal Investigator — Yonsei University
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided